CLINICAL TRIAL: NCT04357041
Title: Effects of Stay-at-home Guidance on Dietary Intake, Physical Activity and Overall Well-being During COVID-19 Public Health Crisis
Brief Title: COVID-19 Survey Study on Dietary Intake, Physical Activity and Overall Well-being
Acronym: CoVS
Status: Completed | Type: Observational
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-2020-91
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: ALL, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research is to collect dietary intake, physical activity, mood and stress data during and after the Illinois shelter-in-place and social distancing orders for the COVID-19 pandemic. The study's intent is to capture data during this unprecedented time to understand the non-infection consequences of social distancing and shelter-in-place, including duration of affect after orders are lifted.

DETAILED DESCRIPTION:
The proposed study is an observational study. The study will include our previous subjects, those who are following the shelter- in- place order due to the COVID-19 pandemic. Demographic data of individuals participating in the study will be recorded. During this 12-month protocol, participants will be contacted through email to complete online questionnaires on weekly basis for 8 weeks, and then once every 4 weeks until the end of the study. Subjects will record their one-day food intake, physical activity, sleep, and stress and anxiety level, which takes ~1 hour to complete.

Subjects will be recruited through our CNRC databases of individuals who come to our clinic in the past 1 year, online advertisement, and word of mouth. A phone and/or email will be administered to ensure their eligibility using our standard tools and protocols. People who are willing and able to participate and meet the basic screening eligibility will be contacted through email for informed consent and the continuing of the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited through our CNRC databases of individuals who come to our clinic in the past years, online advertisement, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Automated Self-Administered 24-Hour Dietary Recall (ASA24) | 0-12 months
  The ASA24 system will be used to document the study participant diet during the study period.
International Physical Activity Questionnaire (IPAQ) | 0-12 months
  IPAQ will be used to evaluate the current physical activity level of the participants during the study period. All continuous scores are expressed in MET-minutes/week, Walking = 3.3 METs, Moderate PA = 4.0 METs and Vigorous PA = 8.0 METs.

SECONDARY OUTCOMES:
Health-Related Quality of Life SF-12 Scale | 0-12 months
  Short Form 12 (Short Form12- SF12) quality of life scale will be used to evaluate health-related quality of life during the study period.The SF-12v2 is a health-related quality-of-life question- naire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vi- tality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). the raw scores could be transformed to provide scores for eight scales, each ranging from 0 (the worst) to 100 (the best)
State trait inventory for cognitive and somatic anxiety (STISA). | 0-12 months
  STISA will be used to measure state and trait anxiety as well as cognitive and somatic anxiety during the study period.scale consists of 21 items that are rated on a 4-point Likert scale. Both the STICSA State and Trait scales were designed to have two factors. One factor reflects the cognitive symptoms of anxiety (10 items, highest score: 40 (the worst), lowest score 10 (the best) ), and the second factor reflects the somatic symptoms of anxiety (11 items, highest score: 44 (the worst), lowest score 11(the best)).
Beck Depression inventory (BDI) | 0-12 months
  BDI will be used to investigate the stress levels of the individuals participating in the study during the study period. The highest possible total for the whole test would be 36, the lowest would be 0. scoring category: 1-10: normal; 11-16 Mild mood disturbance; 17-20: Borderline clinical depression; 21-30
  :Moderate depression; 31-40:Severe depression; over 40: Extreme depression

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States